CLINICAL TRIAL: NCT00003958
Title: Randomized Study of Vincristine, Actinomycin-D, and Cyclophosphamide (VAC) Versus VAC Alternating With Vincristine, Topotecan and Cyclophosphamide for Patients With Intermediate Risk Rhabdomyosarcoma
Brief Title: Combination Chemotherapy in Treating Patients With Previously Untreated Rhabdomyosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9803; NCI-2012-02302 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRS-D9803 (Other: Intergroup Rhabdosarcoma Group); COG-D9803 (Other: Children's Oncology Group); POG-D9803 (Other: Pediatric Oncology Group); CDR0000067157 (Other: Clinical Trials.gov); CCG-D9803 (Other: Children's Cancer Group); U10CA098543 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Adult Malignant Mesenchymoma; Adult Rhabdomyosarcoma; Alveolar Childhood Rhabdomyosarcoma; Childhood Malignant Mesenchymoma; Embryonal Childhood Rhabdomyosarcoma; Embryonal-botryoid Childhood Rhabdomyosarcoma; Nonmetastatic Childhood Soft Tissue Sarcoma; Previously Untreated Childhood Rhabdomyosarcoma; Stage I Adult Soft Tissue Sarcoma; Stage II Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Malignant mesenchymal tumor; Rhabdomyosarcoma; Sarcoma | interventions — Dactinomycin; Vincristine; Cyclophosphamide; Radiotherapy; Radiation; Topotecan; trioctyl phosphine oxide; Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Vincristine sulfate IV once a wk on wks 0-12, 15, 18-24, 27, 30-36, and 39. Dactinomycin IV once a wk on wks 0, 3, 6, 9, 12, 21, 24, 27, 30, 33, 36, and 39. Cyclophosphamide IV once a wk on wks 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, and 39. After 12 weeks of chemotherapy, depending on tumor shrinkage, pts may undergo surgery. After recovery from therapeutic conventional surgery, patients receive radiation therapy once a day, 5 days a wk, during wks 12-18. For pt receiving radiotherapy during wks 0-6, dactinomycin is omitted during wks 3 and 6 and during wks 15 and 18. For patients receiving radiotherapy during wks 12-18, dactinomycin is omitted during wks 15 and 18. Patients with adequate response at wk 24 continue chemotherapy during wks 24-39. All pts receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning 24 hours after completion of each course of chemotherapy and continuing 1 year, until hematopoietic recovery.
  Interventions: Biological: dactinomycin; Drug: vincristine sulfate; Drug: cyclophosphamide; Procedure: therapeutic conventional surgery; Radiation: radiation therapy; Biological: filgrastim; Biological: sargramostim; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive treatment as in arm I, except dactinomycin is replaced with topotecan hydrochloride IV over 15-30 minutes daily for 5 days during weeks 3, 9, 21, 27, 33, and 39.
  All patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning 24 hours after completion of each course of chemotherapy and continuing 1 year, until hematopoietic recovery.
  Interventions: Drug: vincristine sulfate; Drug: cyclophosphamide; Procedure: therapeutic conventional surgery; Radiation: radiation therapy; Drug: topotecan hydrochloride; Biological: filgrastim; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: dactinomycin — Given IV
  Other Names: ACT-D; actinomycin C1; AD; Cosmegen; DACT
  Arms: Arm I
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Procedure: therapeutic conventional surgery — Undergo surgery
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
  Arms: Arm II
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase III trial is comparing two different combination chemotherapy regimens to see how well each works in treating patients with previously untreated rhabdomyosarcoma or sarcoma. Drugs used in chemotherapy, such as dactinomycin, cyclophosphamide, vincristine, and topotecan, use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective in treating rhabdomyosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the early response rates, failure-free survival, and survival of patients with intermediate-risk rhabdomyosarcoma treated with surgery, radiotherapy, and vincristine, dactinomycin, and cyclophosphamide (VAC) vs VAC alternating with vincristine, topotecan, and cyclophosphamide.

II. Compare the acute and late effects of these two treatment regimens in these patients.

III. Determine the rate of second-look surgery in selected patients with bulk residual tumor at diagnosis (i.e., Clinical Group III) and the proportion of these that render the patient tumor free or with microscopic tumor only.

IV. Determine the rate of local failure in selected patients with bulk residual tumors at diagnosis (i.e., Clinical Group III) who, after second-look resection, have response-adjusted radiotherapy dose reduction.

V. Determine if preoperative radiotherapy followed by second-look surgery is feasible for selected patients with bulk residual disease (i.e., Clinical Group III) who respond poorly to induction chemotherapy.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease (embryonal histology, stage II or III, Clinical Group III vs embryonal histology, Clinical Group IV, less than 10 years of age vs alveolar or undifferentiated sarcoma histology, stage I, Clinical Group I vs alveolar or undifferentiated sarcoma histology, stage II or III, Clinical Group II or III). Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive vincristine IV over 5-10 minutes once a week on weeks 0-12, 15, 18-24, 27, 30-36, and 39. Dactinomycin IV is administered over 15-20 minutes once a week on weeks 0, 3, 6, 9, 12, 21, 24, 27, 30, 33, 36, and 39. Cyclophosphamide IV is administered over 30-60 minutes once a week on weeks 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, and 39. After the initial 12 weeks of chemotherapy, depending on tumor shrinkage, patients may undergo surgery. After recovery from surgery, patients receive radiotherapy once a day, 5 days a week, during weeks 12-18. For patients receiving radiotherapy during weeks 0-6, dactinomycin is omitted during weeks 3 and 6 and administered during weeks 15 and 18. For patients receiving radiotherapy during weeks 12-18, dactinomycin is omitted during weeks 15 and 18. Patients showing an adequate response at week 24 continue chemotherapy during weeks 24-39.

Patients with Clinical Group III tumors of a parameningeal site with documented evidence of intracranial extension receive radiotherapy within the first 2 weeks of the initiation of the first course of chemotherapy (day 0).

Patients with Clinical Group II parameningeal tumors and Clinical Group III parameningeal tumors with base of skull erosion and/or cranial nerve palsy without evidence of intracranial extension receive radiotherapy on week 12 (day 84) or immediately thereafter.

Patients with Clinical Group IV parameningeal tumors with distant metastases receive radiotherapy to the primary site on week 12 (day 84). Patients with distant metastases confined to one site may receive radiotherapy to the metastatic site concurrently with therapy to the primary site if it began within 2 weeks of the initiation of chemotherapy (day 0).

Arm II: Patients receive treatment as in arm I, except dactinomycin is replaced with topotecan IV over 15-30 minutes daily for 5 days during weeks 3, 9, 21, 27, 33, and 39.

All patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) subcutaneously beginning 24 hours after completion of each course of chemotherapy and continuing 1 year, until hematopoietic recovery.

Patients are followed every 1-2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven disease of any of the following types:

  * Non metastatic alveolar rhabdomyosarcoma

    * Stage I, II, or III; Clinical Group I, II, or III
  * Stage II or III, Clinical Group III embryonal rhabdomyosarcoma

    * Botryoid
    * Spindle cell
  * Under 10 years, stage IV, Clinical Group IV embryonal rhabdomyosarcoma

    * Botryoid
    * Spindle cell
  * Undifferentiated sarcoma

    * Stage I, II, or III; Clinical Group I, II, or III
  * Ectomesenchymoma

    * Stage I, II, or III; Clinical Group I, II, or III, with alveolar features
    * Under 10 years, Stage IV, Clinical Group IV, with embryonal features
* No more than 6 weeks since initial surgical procedure (e.g., biopsy) giving the definitive diagnosis
* No parameningeal rhabdomyosarcoma with positive CSF cytology or multiple intracranial metastases
* Bilirubin no greater than 1.5 mg/dL
* Creatinine normal* for age
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior chemotherapy
* Prior steroids allowed
* No prior radiotherapy
* See Disease Characteristics

Max Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 702 (Actual)
Dates: Start 2002-09; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Long-term failure-free survival (FFS) between the two treatment groups | Up to 5 years

SECONDARY OUTCOMES:
Overall survival between treatments | Up to 5 years
Rate of second look surgery | Week 12
Proportion of patients rendered tumor-free or with microscopic tumor only | Week 12
Estimation of the rate of local failure for the patients who undergo second look surgery | Week 12
  Done using standard cumulative incidence curves.

CONTACTS AND LOCATIONS:
Overall Officials: Carola Arndt, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States